CLINICAL TRIAL: NCT05937529
Title: Impact of a Cream Containing Madecassoside and 5 % Panthenol in Post Photodynamic Therapy Procedure for Actinic Keratosis: A Randomized, Controlled Trial
Brief Title: Impact of Madecassoside and 5 % Panthenol Cream in Post Photodynamic Therapy for Actinic Keratosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Collaborators: L'Oreal (Industry)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Professor, PhD., dr. med., Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23015740
Record Dates: First submitted 2023-06-08; First posted 2023-07-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — dexpanthenol

STUDY DESIGN:
Intervention Model Description: A randomized, intraindividual controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daylight PDT + Cicaplast (Experimental): Pretreatment with currettage. Metvix cream. Daylight PDT. Application of Cicaplast to test area immediately after dPDT. Cicaplast application twce daily for 14 days.
  Interventions: Other: Cream containing madecassoside and 5 % panthenol; Other: Daylight PDT
- Daylight PDT (Active Comparator): Pretreatment with currettage. Metvix cream. Daylight PDT. No post treatment.
  Interventions: Other: Daylight PDT

INTERVENTIONS:
Other: Cream containing madecassoside and 5 % panthenol — Immediately after daylight PDT, Cicaplast is administrated as post treatment. The patients are instructed to apply the cream twice daily for 14 days.
  Other Names: Cicaplast Baume B5+
  Arms: Daylight PDT + Cicaplast
Other: Daylight PDT — Daylight PDT performed with 2 hours of artifical indoor light.

SUMMARY:
Premalignant AKs are highly frequent in the light-skinned populations with an increasing incidence. PDT is considered a well-establish treatment for these lesions, and therefore it is essential to achieve an optimal and effective treatment as possible. The present study proposes a new post-treatment modality with application of an anti-inflammatory moisturizer Cicaplast Baume B5+ to the treated areas that may improve the overall patient satisfaction and minimize the local skin reactions. Treatment regime consists of two daily applications of Cicaplast Baume B5+ for 14 days, and this regime is not associated with increased risk of systemic AEs or serious events.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. > 18 years of age or older at baseline
3. Fitzpatrick skin type I-III
4. Clinical AKs in two symmetrical areas on the face or on the chest, presented with at least ten AKs
5. Female subjects of childbearing potential must be confirmed not pregnant by negative pregnancy test prior to study inclusion and must use a safe contraceptive method during the study

Exclusion Criteria:

1. Previous exposure to PDT, energy-based devices, or AK treatment on the study areas within 3 months
2. Pregnant or lactating women
3. Patients with known allergy to MAL or any ingredients in Cicaplast, Baume B5+
4. Concomitant treatment with immunosuppressant drugs
5. Infiltrating tumors in the treatment areas
6. Known porphyria
7. Other skin diseases present in the test area at baseline
8. Non-eligibility at the discretion of the investigator (e.g. non-compliance, unavailability or other reasons the subject is not believed to be able to comply with the clinical trial protocol)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Changes in clinically assessed local skin responses after PDT in Cicaplast Baume B5+ treated skin vs. non-post-treated skin from baseline to day 30 | From baseline to day 30
  Clinical evaluation of erythema, edema, and crusting will be done in the two treatment areas at all visits and scored on a four-point scale (0-3): None, mild, moderate, or severe
Evaluation of AK identification and grading before PDT and following PDT treatment in skin treated with Cicaplast Baume B5+ treated skin vs. non-post-treated skin | Evaluated at baseline and at day 30
  Evaluation of clinical response including AK identification and grading will be performed by trained physicians at baseline and at follow-up visits. AK identification and grading will be performed according to Olsen grade classification system:
  * Grade I: Flat, pink maculae without signs of hyperkeratosis and erythema often easier felt than seen
  * Grade II: Moderately thick hyperkeratosis on background of erythema that easily felt and seen
  * Grade III: Very thick hyperkeratosis Occurrence of new AKs in the treatment areas will be recorded at day 30 using the baseline template. The number and severity of the new lesion in the treatment areas will be recorded.
Changes in local skin responses after PDT in Cicaplast Baume B5+ treated skin vs. non-post-treated skin | From baseline to day 30
  OCT system will be used to visualize the epidemis and upper dermis and changes in the cutanous microvascular morphology. All images will be evaluated qualitatively and quantitively using the integrated OCT software.

SECONDARY OUTCOMES:
changes in the skin barrier function from baseline to day 30 | from baseline to day 30
  Skin barrier function is assessed by measurements of trans-epidermal water loss (TEWL) with DermaLab, Cortex Technology, Hadsund, Denmark. Patients will be adjusted to room temperature before TEWL measurements, and skin pH will be measured using a pH-meter from DermaLab, Cortex Technology, Hadsund, Denmark. All measurements will be performed in triplicates and median value will be calculated.
Changes in pigmentation and redness of the skin from baseline to day 30 | From baseline to day 30
  The level of erythema and melanin will be estimated at the treatment areas in the face or the décolleté using the CE-marked Skin Colormeter DSM.
  In addition, erythema and melanin will be estimated in the face using the VISIA, Canfield imaging system, Fairfield, NJ, USA. VISIA uses standard incandescent light, ultraviolet (UV) and cross-polarized light, and generates a series of high-resolution images to determine the patient's overall skin condition. The images will be analyzed with Canfield's software RBX Technology.
Pain during PDT treatment | During the procedure
  Will be evaluated by the patient on a numerical scale 0-10: 0 = none, 10 = worst imaginable pain
Pain in the treatment areas | from day 1 to day 30
  Pain will be evaluated by the patient from day 1 to day 30 by completing a diary with information on pain in the Cicaplast Baume B5+ treated area vs. the non-post-treated area . The scale 0-10: 0 = none, 10 = worst imaginable pain will be used.
Incidence of prutitus in the treatment areas from day 1 to day 30 | from day 1 to day 30
  Patients will be asked to evaluate the incidence of prutitus in Cicaplast Baume B5+ treated area and the non-post-treated area. Pruritus will be evaluted on the scale 0-3: 0 = none, 1 = light, 2 = moderate, 3 = severe
Patients satisfaction with the treatment of daylight PDT + Cicaplast Baume B5+ compared to daylight PDT alone | from baseline to day 30
  Patients will be asked to evaluate their satisfaction with the treatment on a scale 0-10: 0 = could not be more unsatisfied, 10 = could not be more satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, MD PhD DMSc, Principal Investigator — Department of Dermatology Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark